CLINICAL TRIAL: NCT00329342
Title: Return to Work Interventions for Patients With Low Back Pain During Inpatient Rehabilitation: a Quasi-Experimental Study
Brief Title: Return to Work Interventions for Patients With Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Forschungsinstitut für Balneologie und Kurortwissenschaft Bad Elster (Other Government)
Collaborators: European Union (Other); Federal ministry of labour and social affairs (Unknown)
Allocation: Non-Randomized | Model: Parallel | Masking: None
Other Study IDs: RTW-LBP-1
Record Dates: First submitted 2006-05-23; First posted 2006-05-24 (Estimated); Last update posted 2007-11-27 (Estimated); Status verified 2007-11

CONDITIONS: Low Back Pain
Keywords: Low back pain;; Return to work;; Posture
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Behavioral: Occupational ergonomic training
- 2 (No Intervention)

INTERVENTIONS:
Behavioral: Occupational ergonomic training — Adequate postural habits in activities of daily living
  Arms: 1

SUMMARY:
Low back pain has become a major concern to employees and employers because of its negative impact on employee health and productivity.

The objective of this study is to investigate whether a return-to-work intervention conducted during inpatient rehabilitation improves functional limitations that are related with low back pain and interfere with job performance.

DETAILED DESCRIPTION:
In recent years most industrialized nations have been confronted with a dramatic increase in cases dealing with back pain; in Germany, back pain belongs to the major individual and societal health problems with associated costs that have put a strain not only on health care systems. Besides frequent demand for medical services, loss of production (due to temporal sick leave) and disability allowances are important economic factors. In total, the estimated annual costs caused by back pain range between 16 and 22 billion Euros. Population based studies revealed high life-time prevalence with 80% report having ever experienced back pain. The point prevalence lies between 30 and 40%. Approximately one-fourth to one-third of those affected suffer from clinically significant back pain. Epidemiological evidence for the prevalence of back pain, its severity, course and associated risk factors is extensive; however, little systematic knowledge is available about treatment of back pain especially about return-to-work interventions.

This study is designed as a quasi-experimental study to evaluate benefits of return-to-work interventions during medical rehabilitation. Positive effects are expected for low back pain related functional limitations and subsequently job performance. The intervention tested is based on the biomechanical model of chronic pain that assumes a relationship between external strain, body posture, muscle activity, and intravertebral pressure. According to this model, chronic low back pain is partially caused by overexertion and poor postural habits. The intervention aims at lowering the impact of biomechanical stress by training an adequate body posture while performing activities of daily living or job-related activities. Additionally, performing job-related activities target fear-avoidance beliefs especially assumptions about the connection between pain and work activities. The experimental group training good postural habits while performing activities of daily living or job-related activities (additionally to standard rehabilitation activities such as physiotherapy or education and counselling) will be compared with participants receiving a standard rehabilitation only.

Outcome measures are assessed at baseline, post-intervention, and 6 month post-intervention.

ELIGIBILITY:
Inclusion Criteria:

* Chronic low back pain
* Undergoing inpatient rehabilitation
* Working age

Exclusion Criteria:

* Receiving or applying for retirement pension
* Diagnostic findings that require surgery

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2006-04; Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
Low Back Pain Disability: Oswestry Disability Index (ODI) | 6 months

SECONDARY OUTCOMES:
Return-to-work (RTW) outcomes: Duration of time out of work, RTW-status | 6 months
Fear avoidance: Fear-Avoidance Beliefs Questionnaire (FABQ) for Patients with Back Pain | 6 months
Vitality: SF-36 vitality | 6 months
Ergonomic competence: Rating of posture and movement. | 3 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Martina Markes, Principal Investigator — Forschungsinstitut fuer Balneologie und Kurortwissenschaft
Locations (1):
- Vogtlandklinik Bad Elster, Bad Elster, Germany

REFERENCES:
- [Background] Schmidt CO, Kohlmann T. [What do we know about the symptoms of back pain? Epidemiological results on prevalence, incidence, progression and risk factors]. Z Orthop Ihre Grenzgeb. 2005 May-Jun;143(3):292-8. doi: 10.1055/s-2005-836631. German. PMID 15977117
- [Background] Keller S, Herda C, Ridder K, Basler HD. Readiness to adopt adequate postural habits: an application of the Transtheoretical Model in the context of back pain prevention. Patient Educ Couns. 2001 Feb;42(2):175-84. doi: 10.1016/s0738-3991(00)00103-8. PMID 11118783
- [Background] Waddell G, Newton M, Henderson I, Somerville D, Main CJ. A Fear-Avoidance Beliefs Questionnaire (FABQ) and the role of fear-avoidance beliefs in chronic low back pain and disability. Pain. 1993 Feb;52(2):157-168. doi: 10.1016/0304-3959(93)90127-B. PMID 8455963
- [Background] Fairbank JC, Couper J, Davies JB, O'Brien JP. The Oswestry low back pain disability questionnaire. Physiotherapy. 1980 Aug;66(8):271-3. No abstract available. PMID 6450426
- [Background] Pfingsten M, Kroner-Herwig B, Leibing E, Kronshage U, Hildebrandt J. Validation of the German version of the Fear-Avoidance Beliefs Questionnaire (FABQ). Eur J Pain. 2000;4(3):259-66. doi: 10.1053/eujp.2000.0178. PMID 10985869
- [Background] Huppe A, Raspe H. [Efficacy of inpatient rehabilitation for chronic back pain in Germany: a systematic review 1980-2001]. Rehabilitation (Stuttg). 2003 Jun;42(3):143-54. doi: 10.1055/s-2003-40099. German. PMID 12813651